CLINICAL TRIAL: NCT05225662
Title: A Study of the Impact of Radiofrequency Ablation on Left Ventricular Function in Supraventricular Tachyarrhythmias Patient Using Speckle Tracking Echocardiography
Brief Title: Impact of Radiofrequency Ablation on Left Ventricular Function in Supraventricular Tachyarrhythmias Patient Using Speckle Tracking Echocardiography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Tantawy, Principal investigator, Assiut University
Other Study IDs: systolic function, ablation
Record Dates: First submitted 2022-01-14; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Left Ventricular Function, Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: radiofrequency ablation — Mesuring change in Speckle tracking analysis before and after the radiofreqency ablation
  Other Names: speckle tracking

SUMMARY:
In this study, we aimed to evaluate atrial and ventricular function in supraventricular tachyarrhythmia patients before and 3 months after RFA using 2DSTE.

DETAILED DESCRIPTION:
Two-dimensional speckle-tracking echocardiography (2DSTE) is a known technique for the evaluation of myocardial function in many conditions. The longitudinal deformation of the left ventricular (LV) mainly occurs in the subendocardial level which is sensitive to injury and it may be used to identify sub-clinical LV dysfunction in cardiomyopathies. Global longitudinal strain, strain rate (SR), and torsion measurements are very promising to identify patients with mild systolic and diastolic dysfunctions which are not reflected in reduced EF.

Tachyarrhythmias that are persistent and recurrent can lead to LV dysfunction. Dyssynchrony is another mechanism that may cause LV dysfunction, as in the case of Wolf Parkinson Syndrome (WPW ). It might be explained by the "collision" of electric stimuli through the normal atrioventricular conduction system and along the accessory pathway (AP) during the systolic phase. 2DSTE has been used to investigate the characteristics of WPW syndrome and confirm the presence of LV dyssynchrony in this condition.

Lelakowski et al. showed that RFA improves LV systolic and diastolic functions in patients with Atrioventricular Nodal Reentry tachycardia (AVNRT).

Recurrent AVNRT attacks increase atrial pressure, leading to elevated atrial wall stress, which causes negative remodeling and systolic impairment. It has been shown that left atrial(LA) functions improved after Radiofrequency ablation RFA, along with LA volume reduction in atrial fibrillation/flutter patients.

the small number of patients and lacking using advanced accurate techniques lead to currently insufficient data in the literature regarding changes in cardiac function following AVNRT & AVRT ablation and whether LV dyssynchrony is reversible after ablation therapy of AVRT or not.

ELIGIBILITY:
Inclusion Criteria:

- Patients with AVNRT or AVRT undergoing RF ablation

Exclusion Criteria:

* - Patient with bundle blocks
* Coronary artery disease
* Diastolic dysfunction ≥grade 2
* Left ventricular hypertrophy
* Diabetes mellitus
* Chronic renal failure (GFR<45ml\min)
* Moderate to severe valvular heart disease
* Patient with bad echo window

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patient with supraventricular tachyarhythmia undergoing radiofrequency ablation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
left ventricular systolic function | baseline and 3 months later
  assessment of left ventricular systolic function by speckle tracking before and after radiofrequency ablation

REFERENCES:
- [Background] Nagai T, Hamabe A, Arakawa J, Tabata H, Nishioka T. The impact of left ventricular deformation and dyssynchrony on improvement of left ventricular ejection fraction following radiofrequency catheter ablation in Wolff-Parkinson-White syndrome: A comprehensive study by speckle tracking echocardiography. Echocardiography. 2017 Nov;34(11):1610-1616. doi: 10.1111/echo.13691. Epub 2017 Sep 19. PMID 28929532
- [Background] Lelakowski J, Dreher A, Majewski J, Bednarek J, Pasowicz M. [Influence of the treatment of the atrioventricular reentry tachycardia by RF catheter ablation on the left ventricular systolic and diastolic function and exercise capacity]. Wiad Lek. 2009;62(2):71-80. Polish. PMID 20141053